CLINICAL TRIAL: NCT03803982
Title: Deep Neuromuscular Relaxation Optimizing Low-Pressure Bariatric Surgery: A Randomized Controlled Trial
Brief Title: Deep Neuromuscular Relaxation Optimizing Low-Pressure Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Dennis Hong MD, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: low pressure pneumoperitoneum
Record Dates: First submitted 2018-12-19; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: The investigators propose to conduct a double-blind RCT comparing deep neuromuscular blockade to standard blockade during bariatric surgery. Participants will be randomized to one of the two groups in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, surgeons, ward and PACU nurses, research assistants, and surgical house-staff will be blinded to the randomization. The anesthesiologist will be aware of the randomization as this will directly impact the anesthetic delivered to the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Neuromuscular Blockade, Sugammadex (Experimental): All patients will receive anesthetic induction and maintenance as per routine using a combination of propofol, opioids, dexamethasone, and 0.6 mg/kg of rocuronium for induction. Patients will also receive lidocaine 1 mg/kg/hour IV infusion, followed by 3-5 mg of morphine equivalents prior to extubation. Patient monitoring will be according to local practice and consist of electrocardiography, blood pressure, heart rate and bispectral index monitoring. Neuromuscular function will be monitored every 20 minutes using a standardized nerve monitor. After induction and intubation, patients in the Deep Neuromuscular Blockade group (experimental group) will receive additional rocuronium to achieve a NMB blockade of TOF of 0 twitch and maintained at this level until reversal.
  Interventions: Procedure: Deep Neuromuscular Blockade; Drug: Sugammadex
- Standard Anesthetic (No Intervention): Patients in the standard anesthetic (or control group) will also receive anesthetic induction as per routine using a combination of propofol, opioids, dexamethasone, and rocuronium, with a lidocaine infusion. Patient monitoring will be similar to the experimental group, with electrocardiography, blood pressure, heart rate, and bispectral index monitoring. Patients in the control group will receive rocuronium 30 mg intravenous prior to intubation, followed by repeated 10 mg doses to reach a TOF of 1-2 twitches.

INTERVENTIONS:
Procedure: Deep Neuromuscular Blockade — The proposed intervention in this study is delivery of an anesthetic with Deep Neuromuscular Blockage (NMB), which will be defined as a TOF of 0 and 2-3 twitches in the post-tetanic count.
  Arms: Deep Neuromuscular Blockade, Sugammadex
Drug: Sugammadex — Sugammadex will be used to reverse the deep neuromuscular blockade in the experimental group.
  Arms: Deep Neuromuscular Blockade, Sugammadex

SUMMARY:
This study aims to evaluate the use of deep neuromuscular blockade and low-pressure pneumoperitoneum in bariatric surgery. The investigators propose to conduct a double-blind randomized controlled trial (RCT) comparing deep neuromuscular blockade versus standard blockade, and its impact on operative conditions during bariatric surgery. This trial will be conducted at one of the highest volume bariatric centers in Canada. This study also aims to examine the effects of deep neuromuscular blockade on patient-relevant outcomes, including postoperative pain and narcotic use. The investigators anticipate this study will facilitate the continual improvement of care provided to a growing number of bariatric patients.

DETAILED DESCRIPTION:
This will be a double-blind randomized controlled trial comparing patients undergoing a deep neuromuscular blockade with a paralytic reversal agent versus patients undergoing standard anesthetic protocols in low-pressure pneumoperitoneum bariatric surgery. The study population will include patients aged 18-65 referred to St. Joseph's Healthcare for Roux-en-Y Gastric Bypass (RYGB) after completion of standard work-up for bariatric surgery through the Ontario Bariatric Network (OBN). The investigators plan to recruit and randomize 100 patients in a 1:1 ratio between deep NMB and standard anesthetic in low-pressure pneumoperitoneum bariatric surgery. Once enrolled in the study, patients will be assigned to one of the two groups using computer-based randomization on REDCap software. Allocation will be concealed until the time of the operation and will be provided directly to the anesthetist in opaque envelopes. The anesthetist will be aware of the assigned group, but the patient, surgeon, PACU nurses, ward nurses, research assistants and house staff will be blinded. The primary outcomes to be examined will include maximum intra-abdominal pressure, Leiden-Surgical Rating Scale, and postoperative pain scores. Secondary outcomes will include operative time, postoperative nausea, postoperative narcotic use, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets NIH criteria for bariatric surgery and has not received a previous bariatric surgical procedure
* The patient is aged 18-65 years and has completed the screening and preparation process prescribed by the Ontario Bariatric Network

Exclusion Criteria:

* Inability to give informed consent
* ASA > 4
* Planned procedure other than RYGB or contraindications to RYGB
* BMI > 55 kg/m2
* Revisional procedure
* Allergies or suspected allergies to anesthetic medications (rocuronium or sugammadex)
* Renal insufficiency (GFR < 30ml/min)
* Family or personal history of malignant hyperthermia or personal history of neuromuscular disease
* History of chronic pain needing daily medications for the last >3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Maximum IAP | Intraoperatively
  Maximum Intra-Abdominal Pressure, as assessed by the degree of pneumoperitoneum for each position (supine and reverse Trendelenburg)
Leiden-Surgical Rating Scale | Intraoperatively
  Assessment of operating conditions, as assessed by the surgeon, assessed at the beginning of each position change (supine and reverse Trendelenburg). Scale ranges from 1 (extremely poor operating conditions) to 5 (optimal conditions).
Postoperative Pain | Post Operative Day 1
  Postoperative pain as reported by the patient. Pain will be assessed on post operative day 1 at 8 am, noon, and 8pm, and an average pain score will then be calculated for post operative day 1. Pain will be assessed on an 11-point scale ranging from 0 (no pain) to 10 (most pain imaginable)

SECONDARY OUTCOMES:
Operative Time | Intraoperative
  Two operative times will be recorded. The first will be related strictly to the surgery, from time of Veress needle insertion to time of removal of the final port. In addition, total operative time will also be recorded which will include time of induction and reversal of anesthesia
Postoperative Nausea | Postoperative nausea scores will be recorded at 8 am, 2 pm, and 8pm on post operative day 1. Nausea will be measured on an 11-point scale ranging from 0 (no nausea) to 10 (most nausea imaginable).
  Postoperative nausea as reported by the patient
Postoperative Narcotic Use | During index admission, up to one week.
  Amount of narcotic used by the patient postoperative
Length of Stay | During index admission; through study completion, an average of 5 days
  Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD, MSc, Principal Investigator — Centre for Minimal Access Surgery

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared